CLINICAL TRIAL: NCT01421602
Title: A Prospective Observational Study on the Use of a Self Fixating Lightweight Polyester Mesh in Open Inguinal Hernia
Status: Completed | Type: Observational
Sponsor: De La Salle University Medical Center (Other)
Responsible Party: Principal Investigator, Michael M. Lawenko MD, FPCS, Assistant Professor, De La Salle University Medical Center
Other Study IDs: AKMRC-11-001
Record Dates: First submitted 2011-08-22; First posted 2011-08-23 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Hernia, Inguinal
Keywords: Inguinal Hernia; Self-fixating mesh; Progrip; Hernia Recurrence; Mesh, Surgical; Recurrence
MeSH Terms: conditions — Hernia, Inguinal; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will hypothesize that the use of a self fixating lightweight mesh in open inguinal repair is feasible in the Philippine setting. It will result in a comparable recurrence rate as published for the traditional Lichtenstein approach.

DETAILED DESCRIPTION:
The specific aim of this study is to assess the feasibility of using a self fixating lightweight mesh in open inguinal hernia under both under regional and local anesthesia in the Philippines. The primary endpoint of which is to assess the recurrence rate at 2 years (with an interim analysis 1 year after the procedure). Secondary endpoints would be to gather data with regards to postoperative pain, post operative surgical complications, wound healing complications, operating factors (mesh deployment time, total operating time), hernia factors (type and size of inguinal hernia).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Informed consent
* Primary inguinal hernia suitable for open inguinal repair
* Reducible hernia

Exclusion Criteria:

* Incarcerated non reducible hernias
* Bleeding disorders
* Patients below 18 (lower age limit) and above 80 (upper age limit) years old
* Hernia defects of greater than 4 cm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential study subjects will be patients who are:
  18 - 80 years old; Has confirmed with the informed consent; Has a primary inguinal hernia (either unilateral or bilateral) which is reducible and amenable to local or regional hernia repair
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2011-09; Primary Completion 2015-01 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Lawenko, MD, Principal Investigator — De La Salle University Medical Center - Department of Surgery
Locations (1):
- De La Salle University Medical Center, Dasmariñas, Cavite, Philippines

REFERENCES:
- [Result] Chastan P. Tension-free open hernia repair using an innovative self-gripping semi-resorbable mesh. Hernia. 2009 Apr;13(2):137-42. doi: 10.1007/s10029-008-0451-4. Epub 2008 Nov 13. PMID 19005611